CLINICAL TRIAL: NCT00145093
Title: The Effects of Organic Chromium Supplementation on Clinical Parameters of the Metabolic Syndrome, in Patients With Type 2 Diabetes Mellitus. A Randomised, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of Chromium Supplementation on Parameters of the Metabolic Syndrome in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Pharma Nord (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04.0536P
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Chromium; Saccharomyces cerevisiae
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Baker's yeast (Bio Chromium)

SUMMARY:
The purpose of this study is to determine whether chromium (yeast), is effective in improving glycaemic control and insulin resistance.

DETAILED DESCRIPTION:
Setting:

Patients meeting the inclusion and not the exclusion criteria will be sent a letter containing information about the study and that they will be called within 2 weeks by one of the investigators. If the patient agrees to come for a fist visit he or she will be invited for a first visit to come to the general practice of Heerde.

Informed Consent:

During the telephone call and the first visit, patients will be able to ask any question. When the patient is properly informed and gives written informed consent the patient will be included for this study. Specific items such as duration of the study, the frequency of follow-up visits, and the voluntary nature of participation will be discussed prior to obtaining informed consent. Also, because of potential reproductive toxicity (no reports are known of developmental toxicity studies on Cr3+ compounds given orally), we will advice patients to take contraceptive precautions (33).

Stop criteria:

When a patient has any possible drug intolerance the patient will be asked to contact us. We will note every possible side effect. If there is any serious side effect the patient will be asked to stop with the intervention medication.

Power and Sample Size Calculations:

Sample size was calculated by using the computer program G-power. Mean HbA1c of patients with HbA1c 7-8,5% in a general practise in our region is 7,70% (SD 0,44). Powered to detect a 0,5% absolute reduction in HbA1c in the six-month follow-up of patients treated with chromium as compared to placebo patients. With a power 95%, alpha 0.05 2-tailed, the total sample size is 44 (22 in the first group and 22 in the second group).

Randomisation:

60 patients who will meet the inclusion criteria are randomly assigned in a double-blind trial to receive treatment A or B in addition to their current therapy for six months. Method of blinding randomisation: drug packages are labelled with the randomisation code by the hospital pharmacy. Neither the physician nor the patient will be informed of the treatment. There is no delay between study enrolment and randomisation.

Intervention:

Two treatment protocols are proposed. Treatment A consist of 400 microgram Bio-chromium/day and treatment B consists of a placebo. One type of chromium tablets will be made; 100 microgram Cr/tablet. Placebo is made to appear identical with the chromium tablets. Patients are instructed to ingest 2 tablets of the study drug with breakfast and 2 with diner.

Measures:

Medical history consists of duration of diabetes, diabetes medication, general medication, renal or hepatic diseases and recent complaints. Body fat percentages will be measured using the OMRON BF306 (HBF-306-E). Patients are weighed while wearing clothes on bare feet. Length is measured while standing on bare feet and blood pressure measured when the patient is in a sitting position according to the Dutch College of General Practitioners (34).

Serum creatinine, hepatic enzyme (PT), HbA1c, Haemoglobin (Hb), fasting glucose, fasting insulin, serum total cholesterol, LDL, HDL, and triglycerides will be measured at baseline with the standard procedure in our hospital (Weezenlanden Location, Isala Clinics).

At baseline and after six months, also serum chromium will be measured. Extra citrate and serum collection tubes will be frozen for additional measurements, when needed. Also 24-h urine will be collected at baseline and after 6 months and volume, creatinine, protein and albumin will be measured. Three tubes containing both 2 cc of urine will be frozen for additional measurements. These (extra) analyses will only be made after given information and approval of the patient, and after approval of the medical ethical committee.

Follow up:

At baseline, an appointment will be made for the following visit and an appointment for a telephone call after 4 weeks. During this call, patients will be asked if they had any complaint which started after inclusion to this study. For stimulating compliance, patients will be asked how they use their tablets. When this is different from described in this protocol, patients will be advised accordingly. Furthermore, patients will be able to ask any question during this telephone call.

Patients can call us when there is any possible adverse or toxic effects of the drug during office hours.

After 3 months, only HbA1c and Hb will be measured. The other measures as described above, except for length will be measured at baseline and after 6 months.

Handling of losses to follow-up:

Patients withdrawn from study medication will receive regular follow-up until the end of the 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with haemoglobin A1c level between 7 and 8.5% at the last visit
* treated with oral blood glucose lowering therapy, which has not been changed for the last three months.

Exclusion Criteria:

* pregnant women; women trying to become pregnant
* patients with a serum creatinine concentration over 150 micromol/l in men and 120 micromol/l in women, Cockcroft < 50 ml/min
* hepatic enzyme levels (ALAT) over 90 U/l (2 x upper limit)
* patients known with allergy or intolerance for yeast
* patients currently taking chromium supplements
* patients treated with insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2005-02

PRIMARY OUTCOMES:
To determine the effect of Baker's yeast treatment on glycemicic control and insulin resistance when given in combination with oral blood glucose lowering therapy to patients with type 2 diabetes mellitus

SECONDARY OUTCOMES:
To determine the effect of Baker's yeast treatment on serum lipids, blood pressure, body fat percentage and BMI when given in combination with oral blood glucose lowering therapy to patients with type 2 diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Henk JG Bilo, MD PhD FRCP, Principal Investigator — Isala clinics, medical research foundation
Locations (1):
- General Practice, Heerde, Netherlands